CLINICAL TRIAL: NCT04986982
Title: Randomised, Double-blind, Placebo-controlled, Clinical Study to Evaluate the Effect of Opicapone 50 mg on Parkinson's Disease Patients With End-of-dose Motor Fluctuations and Associated Pain.
Brief Title: OpiCapone Effect on Motor Fluctuations and pAiN
Acronym: OCEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-91067-404; 2020-001175-32 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opicapone 50 mg (Experimental): Opicapone (BIA 9-1067)
  Interventions: Drug: Opicapone 50 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Opicapone 50 mg — Opicapone (BIA 9-1067) 50 mg hard capsules. Oral administration, once daily, at least 1 hour before or after the last daily dose of L-dopa/DDCI
  Other Names: BIA 9-1067
  Arms: Opicapone 50 mg
Other: Placebo — Matching placebo hard capsules. Oral administration, once daily, at least 1 hour before or after the last daily dose of L-dopa/DDCI
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy of 50 mg opicapone when administered with the existing treatment of levodopa (L-dopa) plus a dopa decarboxylase inhibitor (DDCI), in Parkinson's disease (PD) patients with end-of-dose motor fluctuations and associated pain

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multi-centre, parallel group, interventional clinical study in PD patients with end-of-dose motor fluctuations and associated pain. The study consists of a 1-week screening period, a 24-week double-blind treatment period and 2 weeks of follow-up period. The duration of treatment for the individual patient is expected to be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form and to comply with all aspects of the study.
2. Male or female patients aged 30 years or older.
3. Experiencing PD associated pain for at least 4 weeks prior to V1.
4. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (2006) or according to MDS Clinical Diagnostic Criteria (2015).
5. Disease severity Stages I-III (modified Hoehn & Yahr staging) at ON.
6. Treated with 3 to 8 intakes per day of L-dopa/DDCI (which may include a slow-release formulation), on a stable regimen for at least 4 weeks before V1.
7. In case of any other anti-PD-treatment, it should be on a stable regimen for at least 4 weeks before V1, and not likely to need any adjustment until V6.
8. No changes in chronic treatment regimen for pain within the last 4 weeks before V1. This includes medication (including but not limited to paracetamol, opioids, nonsteroidal anti-inflammatory drugs [NSAIDS], antidepressants, anticonvulsants and corticosteroids) and non-medication therapies (including but not limited to transcutaneous electrical nerve stimulation and bioelectrical therapy).
9. Signs of "wearing-off" phenomenon (end-of-dose motor fluctuations) with average total daily OFF time while awake of at least 1.5 hours, excluding the early morning pre-first dose OFF, despite optimal anti-PD therapy (based on investigator's assessment).
10. Domain 3 of KPPS ≥ 12.
11. For females: Postmenopausal for at least 2 years before V1, surgically sterile for at least 6 months before V1, or practicing effective contraception until V6. Female patients who request to continue with oral contraceptives must be willing to use non-hormonal methods of contraception in addition during the course of this study.

    For males: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception during the treatment period until V6.
12. Have filled-in self-rating diary in accordance with the diary instructions and with ≤ 3 missing entries per day, in the 3 days preceding V2a/V2b.
13. With at least 1.5 OFF hours per day, excluding the early morning pre-first dose OFF period (i.e. the time between wake-up and response to the first L dopa/DDCI dosage), as recorded in at least 2 of the 3 days in the self-rating diary for the 3 days preceding V2a/V2b.
14. Results of the screening laboratory tests are considered acceptable by the investigator (i.e. not clinically relevant for the well-being of the patient or for the purpose of the study).
15. Domain 3 of KPPS ≥ 12.
16. Adequate compliance to relevant (PD and pain related) concomitant medication during the screening period (based on the investigator's judgment).

Exclusion Criteria:

1. Non-idiopathic PD (atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
2. Severe and/or unpredictable OFF periods, according to investigator judgement.
3. Major/prominent non-PD-related pain (e.g. due to malignant disease).
4. Treatment with prohibited medication: entacapone, tolcapone, monoamine oxidase (MAO) inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation, rasagiline up to 1 mg/day or safinamide up to 100 mg/day), or antiemetics with antidopaminergic action (except domperidone) within the last 4 weeks before V1.
5. Previous or planned (during the entire study duration) L-dopa/carbidopa intestinal gel infusion, deep brain stimulation or stereotactic surgery (e.g. pallidotomy, thalamotomy).
6. Treatment with apomorphine within the last 4 weeks before V1 or likely to be needed at any time until V6.
7. Previous or current use of opicapone.
8. Use of any other IP, currently or within the 3 months (or within 5 half-lives of the IP, whichever is longer) before V1.
9. Past (within the past year) or present history of suicidal ideation or suicide attempts.
10. Current or previous (within the past year) alcohol or substance abuse excluding caffeine or nicotine.
11. Phaeochromocytoma, paraganglioma, or other catecholamine secreting neoplasms.
12. Known hypersensitivity to the excipients of IP (including lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption) or of rescue medication.
13. History of neuroleptic malignant syndrome or non-traumatic rhabdomyolysis.
14. History of severe hepatic impairment (Child-Pugh Class C).
15. Previous history of psychosis or psychiatric disorders, including severe major depression.
16. Any medical condition that might place the patient at increased risk or interfere with assessments.
17. For females: Pregnant or breastfeeding.
18. Employees of the investigator, study centre, sponsor, clinical research organisation and study consultants, when employees are directly involved in this study or other studies under the direction of this investigator or study centre, and their family members.
19. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kallol Ray Chaudhuri, MD, DSc, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- The Maurice Wohl Clinical Neuroscience Institute - King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: King's Parkinson's Disease Pain Scale — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6174437/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 144 patients were enrolled and 19 patients prematurely terminated the trial.
Period: Overall Study
Arm/Group | Opicapone 50 mg | Placebo
Started | 64 | 63
Safety Set | 64 | 63
Full Analysis Set | 59 | 63
Completed | 53 | 55
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Ineligibility | 3 | 0
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor's discretion | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 122 (96.1%) patients met the criteria for the full analysis set (FAS) including 59 (92.2%) opicapone 50 mg and 63 (100.0%) placebo patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opicapone 50 mg | Placebo | Total
Number analyzed (Participants) | 59 | 63 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.14) | 65.5 (9.39) | 66.2 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 32 | 32 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 59 | 62 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 11 | 17
  Germany | 2 | 5 | 7
  Poland | 14 | 14 | 28
  Italy | 9 | 1 | 10
  Portugal | 7 | 11 | 18
  Czechia | 16 | 10 | 26
  Spain | 5 | 11 | 16
Age, Categorical [Count of Participants; unit: Participants]
  ≥ 18 years - < 65 years | 21 | 29 | 50
  ≥ 65 years - < 85 years | 37 | 34 | 71
  ≥ 85 years | 1 | 0 | 1
Childbearing potential [Count of Participants; unit: Participants] — Population: For childbearing potential, the percentage is based on the number of females.
  Participants
    Yes: number analyzed (Participants) | 27 | 31 | 58
    Yes | 1 | 2 | 3
    No: number analyzed (Participants) | 27 | 31 | 58
    No | 26 | 29 | 55
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.16 (4.934) | 29.10 (5.079) | 28.65 (5.011)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Domain 3 (Fluctuation-related Pain) of KING's PARKINSON's DISEASE PAIN SCALE (KPPS)
Description: The KING's PARKINSON's DISEASE PAIN SCALE (KPPS) evaluates the burden (global and bedside) and characterises various phenotypes of pain in Parkinson's disease. The investigator will complete the questionnaire by interviewing the patient about seven domains and answering to 14 items. The questionnaire will be fill out on Visit 1, Visit 2b/Baseline, Visit 4, Visit 5 and Visit 6/EDV Domain 3 assesses fluctuation-related pain (score range: 0 - 36). Higher score values indicate higher levels of pain.
Time Frame: The questionnaire will be fill out on Visit 1 (Day -7 ±2), Visit 2b/Baseline (Day 1), Visit 4 (Day 29 (±2)), Visit 5 (Day 85 (±4)) and Visit 6/Early Discontinuation Visit (EDV) (Day 169 (±4)) - Up to 24 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opicapone 50 mg | Placebo
Number analyzed (Participants) | 59 | 63
score on a scale
  Visit 1 (Day -7 ±2) | 17.2 (5.72) | 16.7 (5.18)
  Visit 2b (Day 1) | 17.1 (5.58) | 16.9 (5.20)
  Baseline (Day 1) | 17.1 (5.58) | 16.9 (5.20)
  Visit 4 (Day 29 (±2)) - Observed Value | 10.5 (7.92) | 11.0 (7.51)
  Visit 4 (Day 29 (±2)) - Change from Baseline | -6.6 (7.28) | -5.9 (6.02)
  Visit 5 (Day 85 (±4)) - Observed Value | 8.3 (7.27) | 9.3 (5.73)
  Visit 5 (Day 85 (±4)) - Change from Baseline | -8.7 (6.68) | -7.6 (6.13)
  Visit 6 (Day 169 (±4)) - Observed Value | 8.4 (6.93) | 7.5 (6.48)
  Visit 6 (Day 169 (±4)) - Change from Baseline | -8.8 (6.85) | -9.3 (6.24)

ADVERSE EVENTS:
Time Frame: The period of monitored/assessed for the collection of AEs were through study completion, about 3 years.
Arm/Group | Opicapone 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 4/64 | 2/63
Other Adverse Events (participants affected / at risk) | 40/64 | 36/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opicapone 50 mg (N=64) | Placebo (N=63)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opicapone 50 mg (N=64) | Placebo (N=63)
Dyskinesia (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 3 (3)
Parkinson's disease (Nervous system disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4)
On and off phenomenon (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Bradykinesia (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Freezing phenomenon (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (3) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (6) | 3 (3)
Fatigue (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Application site irritation (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (7) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04986982/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04986982/SAP_001.pdf